CLINICAL TRIAL: NCT04833491
Title: Study of the Correlation Between Preoperative Precise Biometrics, Spatial Assessment and Postoperative Visual Quality in Cataract Patients
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: xuwen2021-0189
Record Dates: First submitted 2021-04-02; First posted 2021-04-06 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-03

CONDITIONS: Recruitment of Participants
Keywords: refractive cataract surgery; intraocular lens

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Senile cataract
- Traumatic cataract
- Congenital cataract
- Lens dislocation group
- Complicated cataract

SUMMARY:
This study summarizes the experience of precision treatment and postoperative management of various types of cataract, and intend to further improve the quality of Clinical Cataract diagnosis and treatment.

DETAILED DESCRIPTION:
Based on the existing cataract surgery methods, through prospective follow-up study, this study summarizes the experience of precision treatment and postoperative management of various types of cataract, and intends to further improve the quality of Clinical Cataract diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with monocular or binocular cataract, lens opacity or abnormal position, need surgery

Exclusion Criteria:

* The history of systemic diseases and medication affecting vision, diabetic patients with systemic conditions complicated with retinopathy, uncontrolled blood glucose, severe eye diseases, eye trauma, eye surgery, severe dry eye and ocular surface diseases, strabismus and amblyopia were identified

Ages: 2 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cataract surgery was performed in ophthalmic hospital affiliated to Medical College of Zhejiang University
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | 1 week postoperatively
  The BCVA was measured by the same optometrist at each visit
Best Corrected Visual Acuity | 1 month postoperatively
  The BCVA was measured by the same optometrist at each visit
Best Corrected Visual Acuity | 3 months postoperatively
  The BCVA was measured by the same optometrist at each visit
Uncorrected distance visual acuity | 1 week postoperatively
  The UCVA was measured by the same optometrist at each visit
Uncorrected distance visual acuity | 1 month postoperatively
  The UCVA was measured by the same optometrist at each visit
Uncorrected distance visual acuity | 3 months postoperatively
  The UCVA was measured by the same optometrist at each visit
Intraocular pressure | 1 week postoperatively
  Intraocular pressure measured using non-contact tonometer
Intraocular pressure | 1 month postoperatively
  Intraocular pressure measured using non-contact tonometer
Intraocular pressure | 3 months postoperatively
  Intraocular pressure measured using non-contact tonometer
Tear Breakup Time | 1 week postoperatively
  Tear Breakup Time was performed to assess tear film stability
Tear Breakup Time | 1 month postoperatively
  Tear Breakup Time was performed to assess tear film stability
Tear Breakup Time | 3 months postoperatively
  Tear Breakup Time was performed to assess tear film stability
Endothelial cell density | 1 month postoperatively
  Endothelial cell density was measured by specular microscopy
Contrast sensitivity | 1 month postoperatively
  The contrast sensitivity was recorded in dark environment, glare dark environment, light environment, glare light environment
Defocusing curve | 1 month postoperatively
  From +2.00d to -4.00d, 13 different diopter states were obtained by decreasing the spherical lens degree of +0.50d, and the defocus curve was formed
Stereoscopic vision | 1 month postoperatively
  The binocular diopter was not corrected. The stereopsis test card was used to record the arc seconds of random points, animals and circles
Glasses usage frequency | 3 months postoperatively
  The frequency of long / medium / short distance use of corrective glasses was scored as 0%, 25%, 50%, 75% and 100%
Optical visual quality questionnaire | 3 months postoperatively
  Glare, halos, starburst and other visual quality problems were graded as mild（1 score), moderate（2 score) and severe（3 score)
Visual satisfaction | 3 months postoperatively
  The visual acuity satisfaction of distance / middle / near distance was scored from 0 (totally dissatisfied) to 10 (totally satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, China

REFERENCES:
- [Derived] Fang J, Shi C, Ma X, Sheng S, Xu J, Zhu S, Feng Y, Zhang Y, Liu L, Zhao H, Xu Z, Xu W. Anterior segment characteristics and spatial variations of different crystalline lens diseases. Photodiagnosis Photodyn Ther. 2025 Aug;54:104693. doi: 10.1016/j.pdpdt.2025.104693. Epub 2025 Jun 26. PMID 40581199
- [Derived] Xu Z, Wang J, Shi C, Ni S, Xu J, Zhu S, Fang J, Xu W. Clinical outcomes of plate-haptic diffractive multifocal toric IOL in cataract eyes with long axial length and corneal astigmatism. Sci Rep. 2025 Apr 7;15(1):11881. doi: 10.1038/s41598-025-97040-0. PMID 40195538